CLINICAL TRIAL: NCT01571141
Title: Polyhexamethylene Biguanide Increases the Regression Rate of Human Papillomavirus (HPV) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: PHMB_HPV
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2011-06

CONDITIONS: HPV Infection
Keywords: HPV; polyhexamethylene biguanide; intraepithelial lesions; regression rate
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monogin (Experimental)
  Interventions: Device: Monogin
- No intervention (No Intervention)

INTERVENTIONS:
Device: Monogin — Gynaecological solution with polyhexamethylene biguanide, pH 4.0
  Arms: Monogin

SUMMARY:
Human papillomavirus (HPV) infection is a worldwide problem strictly linked to the development of cervical cancer. Persistence of the infection is one of the main factors responsible for the invasive progression and women diagnosed with intraepithelial squamous lesions are referred for further assessment and surgical treatments which are prone to complications. Despite this, there are several reports on the spontaneous regression of the infection.

In this study the investigators will evaluate the effectiveness of a long term polyhexamethylene biguanide (PHMB)-based local treatment in improve the viral clearance reducing the time exposure to the infection and avoiding the complications associated with the invasive treatments currently available.

Women diagnosed with HPV infection were randomly assigned to receive six months of treatment with a PHMB-based gynaecological solution (Monogin®) or to remain untreated for the same period of time.

The administration of Monogin® has been performed every three days for fifteen days and then every fifteen days for the subsequent six months.

ELIGIBILITY:
Inclusion Criteria:

* pathologic Pap smear
* positive "high risk" HPV DNA test
* positive colposcopy examination

Exclusion Criteria:

* patients who had undergone wart therapy in the previous six months
* pregnancy
* invasive disease
* immunosuppression
* previous HPV vaccination

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Number of patients with no HPV infection

CONTACTS AND LOCATIONS:
Locations (1):
- Consultorio Familiare Terme Vigliatore, A.S.P. 5, Messina, Italy

REFERENCES:
- [Background] Zanotti KM, Belinson J. Update on the diagnosis and treatment of human papillomavirus infection. Cleve Clin J Med. 2002 Dec;69(12):948, 951-5, 956 passim. doi: 10.3949/ccjm.69.12.948. PMID 12546268
- [Background] Hubner NO, Kramer A. Review on the efficacy, safety and clinical applications of polihexanide, a modern wound antiseptic. Skin Pharmacol Physiol. 2010;23 Suppl:17-27. doi: 10.1159/000318264. Epub 2010 Sep 8. PMID 20829658
- [Background] Marelli G, Papaleo E, Origoni M, Caputo L, Ferrari A. Polyhexamethylene biguanide for treatment of external genital warts: a prospective, double-blind, randomized study. Eur Rev Med Pharmacol Sci. 2005 Nov-Dec;9(6):369-72. PMID 16479742
- [Derived] Gentile A, Gerli S, Di Renzo GC. A new non-invasive approach based on polyhexamethylene biguanide increases the regression rate of HPV infection. BMC Clin Pathol. 2012 Sep 25;12:17. doi: 10.1186/1472-6890-12-17. PMID 23009652